CLINICAL TRIAL: NCT04616924
Title: Study of RHB-204 for the Treatment of Pulmonary Mycobacterium Avium Complex (MAC) Disease in Adults With Nodular Bronchiectasis (CleaR-MAC Trial)
Brief Title: RHB-204 for the Treatment of Pulmonary Mycobacterium Avium Complex Disease
Acronym: CleaR-MAC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: extremely slow enrollment into study
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHB-204-01
Record Dates: First submitted 2020-10-19; First posted 2020-11-05 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2023-06

CONDITIONS: Pulmonary Mycobacterium Avium Complex Infection; Bronchiectasis; Lung Diseases
Keywords: MAC; Bronchiectasis; NTM
MeSH Terms: conditions — Bronchiectasis; Lung Diseases | interventions — Clarithromycin; Rifabutin; Clofazimine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RHB-204 (Experimental): Each capsule contains clarithromycin 158.3mg; rifabutin 40mg; clofazimine 13.3mg.
  Interventions: Drug: RHB-204
- Placebo (Placebo Comparator): Matching placebo will contain riboflavin, a type of B vitamin, which may discolor urine in a similar fashion as RHB-204.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RHB-204 — RHB-204
  Other Names: Clarithromycin 158.3mg, Rifabutin 40mg and Clofazimine 13.3mg
  Arms: RHB-204
Drug: Placebo — Matching placebo to RHB-204
  Arms: Placebo

SUMMARY:
A 2-part multi-center, Phase 3, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of RHB-204 in adult subjects with underlying nodular bronchiectasis and documented MAC lung infection.

DETAILED DESCRIPTION:
A 2-part multi-center, Phase 3, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of RHB-204 in adult subjects with underlying nodular bronchiectasis and documented MAC lung infection.

The co-primary efficacy endpoints at the end of Part 1 evaluate the proportion of patients with sputum culture conversion after 6 months of treatment defined as three consecutive monthly negative sputum cultures at Months 4, 5, and 6 for RHB-204 compared to placebo and the mean change in the Quality of Life Questionnaire - Bronchiectasis (QoL-B) Respiratory Symptoms domain score from baseline to Month 6 for RHB-204 compared to placebo.

At the Month 6 visit (end of Part 1), after all assessments including questionnaires and sputum samples have been collected, subjects will enter Part 2 of the study and receive open-label RHB-204.

In order to comply with current treatment duration guidelines (Nontuberculous Mycobacterial Pulmonary Disease Caused by Mycobacterium avium Complex: Developing Drugs for Treatment - FDA Draft Guidance September 2021) in this protocol subjects will receive active treatment for 12 months after sputum culture conversion. As such, each subject's first negative culture that defines conversion will determine the total duration of their active study drug treatment. The longest duration of active study drug treatment will be 16 months. At the end of study treatment, all subjects will enter a 3-month post-treatment follow-up period (see study design section below for additional details).

To maintain the blind and integrity of the data, an independent team (Sputum Culture Monitors) will inform sites on each subject's treatment duration based on sputum culture conversion. Sputum Culture Monitors will also have access to randomized treatment allocation. All other study related personnel will remain blinded to sputum culture results and treatment allocation (Sponsor, CRO, medical monitors, safety, ECG and sputum laboratories, site personnel as well as participating subjects).

During Part 1, subjects who have completed at least the first 3 months of treatment with study drug, and at the Investigator's discretion, require rescue therapy (alternative anti-NTM treatment) will discontinue study drug (performing an EOT visit) and remain in the study to complete all scheduled study visits and assessments/procedures to Month 6 (performing an EOS visit).

Subjects who complete treatment based on the timeline provided by the Sputum Culture Monitors (EOT visit) and have an ongoing negative sputum culture will be reconsented to enter a follow-up Extension Study, to evaluate sputum culture results at two (2) further time points: 6 months and 12 months following end of treatment (EOT) for each subject in protocol RHB-204-01.

ELIGIBILITY:
Key Inclusion Criteria

* Males and females aged ≥18 years to ≤85 years of age, inclusively
* Have a MAC lung infection documented by one MAC positive culture within 18 months prior to screening and a MAC positive culture at screening (cultures need to be at least 1 month apart). Prior sputum for culture may be obtained from sputum or bronchial washings however, sputum collected during screening must be either spontaneously expectorated by the patient or after sputum induction.
* Have MAC lung infection with evidence of underlying nodular infiltrates and/or bronchiectasis on a chest computed tomography (Chest CT) within 6 months of screening.
* Have symptoms of MAC lung infection that include one of the following: respiratory symptoms such as chronic cough, excessive mucous production, fatigue, dyspnea, hemoptysis or systemic symptoms such as fever, night sweats or loss of appetite.
* Be treatment naïve, or if previously treated for MAC, have not received treatment within the 6 months prior to screening
* Subject's weight is above 41 Kilograms or 90 pounds.

Key Exclusion Criteria

* Cavitary lung disease as observed on a chest CT scan (cavitary lesions exceeding 2 cm in diameter).
* Currently taking or treated in the 6 months prior to screening with any of the following: bedaquiline, clofazimine or any component of American Thoracic Society(ATS)/Infectious Diseases Society of America (IDSA) multi-drug recommended therapy (macrolides, ethambutol, rifabutins/rifampins) for MAC or other multi-drug regime for NTM lung disease
* Clarithromycin minimum inhibitory concentration (MIC) ≥32μg/mL on MAC isolates in screening sputum
* Known hypersensitivity or suspected history of hypersensitivity reactions to clarithromycin, rifabutin, or clofazimine or other drugs in each class
* Subjects requiring chronic supplemental oxygen use (including intermittent or continuous use)
* Planned lung resection surgery for MAC lung disease
* Subjects with Cystic Fibrosis, prior solid organ or hematologic transplant
* Current usage of inhaled products containing amikacin, tobramycin or gentamicin
* History of ventricular arrhythmias or family history of Long QT syndrome, including torsades de pointes
* Corrected QT (QTc) interval on electrocardiogram (ECG) >460 ms for females or >450 ms for males, calculated using Fridericia's formula (QTcF)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Quality of Life Questionnaire - Bronchiectasis (QoL B) Respiratory Symptoms domain score from baseline to Month 6 for RHB-204 compared to placebo | 6 months
  The mean change in the Quality of Life Questionnaire - Bronchiectasis (QoL B) Respiratory Symptoms domain score from baseline to Month 6 for RHB-204 compared to placebo
Sputum culture conversion (SCC) | 6 months
  The proportion of subjects who achieve SCC by Month 6, defined by 3 consecutive monthly negative sputum cultures, without reversion, at Months 4, 5 & 6 for THB-204 compared to placebo.

SECONDARY OUTCOMES:
Part 1 Secondary efficacy objective - Reduction of fatigue | 6 months
  The mean change in the PROMIS Fatigue SF 8a score from baseline to Month 6 for RHB-204 compared to placebo. The PROMIS Fatigue SF 8a score from baseline to Month 6 for RHB-204 compared to placebo.
Part 1 Secondary efficacy objective - Time to culture conversion | 6 months
  The time to SCC (month of first negative sputum culture) for RHB-204 compared to placebo.
Part 1 Secondary efficacy objective - Improvement in Physical Functioning | 6 months
  The mean change in the Short Form 36 Physical Functioning domain score from baseline to Month 6 for RHB-204 compared to placebo.
Part 2 Secondary efficacy objective - Durable Sputum culture conversion at end of study | 19 months
  The proportion of subjects with SCC by Month 6 who sustain negative sputum cultures at Month 16 and negative sputum culture at Month 19 (3 months off treatment) for RHB-204 compared to placebo (durable responders).
Part 2 Secondary efficacy objective - Durable Sputum culture conversion at end of treatment | 16 months
  Measure the proportion of subjects with SCC by Month 6 who sustain negative sputum cultures at Month 16 for RHB-204 compared to placebo.
QoL B Respiratory Symptoms domain score mean change from baseline to Month 16 | 16 months
  The mean change in Quality of Life Questionnaire - Bronchiectasis (QoL-B) Respiratory Symptoms domain scores from baseline to Month 16 for ex-RHB-204 compared to ex-placebo
Part 2 Secondary efficacy objective - Improvement in Quality of Life - Fatigue 16 months | 16 months
  The mean change in the PROMIS Fatigue SF 8a score from baseline to Month 16 for ex-RHB-204 compared to ex-placebo
Part 2 Secondary efficacy objective - Improvement in Quality of Life - Fatigue 19 Months | 19 months
  The mean change in the PROMIS Fatigue SF 8a score from baseline to Month 19 for ex-RHB-204 compared to ex-placebo
Part 2 Secondary efficacy objective - Quality of Life Physical Functioning Symptoms 16 Months | 16 months
  The mean change in the Short Form 36 Physical Functioning domain score from baseline to Month 16 for ex-RHB-204 compared to ex-placebo
Part 2 Secondary efficacy objective - Quality of Life Physical Functioning Symptoms 19 Months | 19 Months
  The mean change in the Short Form 36 Physical Functioning domain score from baseline to Month 19 for ex-RHB-204 compared to ex-placebo
QoL-B Respiratory Symptoms domain scores at Month 19 | 19 Months
  The mean change in Quality of Life Questionnaire - Bronchiectasis (QoL-B) Respiratory Symptoms domain scores from baseline to Month 19 for ex-RHB-204 compared to ex-placebo

CONTACTS AND LOCATIONS:
Overall Officials: Kevin L. Winthrop, MD, MPH, Study Director — Oregon Health and Science University; June L Almenoff, MD, PhD, Study Chair — RedHill Biopharma, Inc.
Locations (25):
- United States (25):
  - Medical Facility, Glendale, California
  - Medical Facility, Palm Springs, California
  - Medical Facility, Farmington, Connecticut
  - Medical Facility, Washington D.C., District of Columbia
  - Medical Facility, Clearwater, Florida
  - Medical Facility, Gainesville, Florida
  - Medical Facility, Margate, Florida
  - Medical Facility 1, Orlando, Florida
  - Medical Facility 2, Orlando, Florida
  - Medical Facility, Sebring, Florida
  - Medical Facility, Vero Beach, Florida
  - Medical Facility, Atlanta, Georgia
  - Medical Facility, Valdosta, Georgia
  - Medical Facility, Kansas City, Kansas
  - Medical Facility, New Orleans, Louisiana
  - Medical Facility, Boston, Massachusetts
  - Medical Facility, Rochester, Minnesota
  - Medical Facility, St Louis, Missouri
  - Medical Facility, Newark, New Jersey
  - Medical Facility, New York, New York
  - Medical Facility, Winston-Salem, North Carolina
  - Medical Facility, Portland, Oregon
  - Medical Facility, Charleston, South Carolina
  - Medical Facility, Tyler, Texas
  - Medical Facility, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: No